CLINICAL TRIAL: NCT02081261
Title: Predicting Acute Kidney Injury After Coronary Artery Bypass Graft : a Simplified Clinical Risk Scoring Model
Brief Title: Predicting Acute Kidney Injury After Coronary Artery Bypass Graft
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, WonHo Kim, Assistant Professor, Samsung Medical Center
Other Study IDs: 2013-12-116
Record Dates: First submitted 2014-03-05; First posted 2014-03-07 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-06

CONDITIONS: Coronary Artery Bypass Surgery; Acute Kidney Injury; Creatinine; Mortality
Keywords: coronary artery bypass surgery; acute kidney injury; creatinine; mortality
MeSH Terms: conditions — Acute Kidney Injury | interventions — Coronary Artery Bypass

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Coronary artery bypass surgery: patients who underwent coronary artery bypass surgery between 2010 and 2012 in Samsung Medical Center
  Interventions: Procedure: Coronary artery bypass surgery

INTERVENTIONS:
Procedure: Coronary artery bypass surgery — coronary artery bypass surgery

SUMMARY:
Acute kidney injury after cardiac surgery is a major complication after cardiac surgery and has been reported to be associated with adverse outcome. There have been many studies reporting risk factor of acute kidney injury after cardiac surgery, but the influence of perioperative variables related to anesthesia and perioperative medication has not been evaluated fully. The investigators attempt to evaluate the influence of perioperative clinical variables including preoperative medication, preoperative albumin level, uric acid concentration, anesthesia technique, use of hydroxyethyl starch, blood glucose level, intraoperative medication, perioperative cardiac function (systolic and diastolic function) and hemodynamic variables during surgery on the incidence of acute kidney injury after coronary artery bypass graft.

DETAILED DESCRIPTION:
Acute kidney injury (AKI) after cardiac surgery is a major complication after cardiac surgery and has been reported to be associated with adverse outcome. There have been many studies reporting risk factor of acute kidney injury after cardiac surgery, but the influence of perioperative variables related to anesthesia and perioperative medication has not been evaluated fully. The investigators attempt to evaluate the influence of preoperative medication, preoperative albumin level, uric acid concentration, NL ratio, anesthesia technique, use of hydroxyethyl starch, blood glucose level, intraoperative medication, perioperative cardiac function (systolic and diastolic) and hemodynamic variables during surgery on the incidence of acute kidney injury after coronary artery bypass graft. Preoperative and postoperative diastolic dysfunction may be associated with postoperative AKI. In addition, preoperative neutrophil-lymphocyte ratio (NLR) which has been reported to be a marked for systemic inflammation and was associated with prognosis in cardiac patients undergoing coronary artery bypass graft or percutaneous coronary intervention. This preoperative or immediate postoperative NLR might be able to predict AKI after coronary artery bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent coronary artery bypass surgery during between 2010 and 2012 in Samsung Medical Center

Exclusion Criteria:

* lack of postoperative creatinine or urine output data
* patients who expired within 24hours after surgery

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who underwent coronary artery bypass surgery during between 2010 and 2012 in Samsung Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 877 (Actual)
Dates: Start 2014-01; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Acute kidney injury diagnosis defined by KDIGO criteria | during 7 days after surgery
  Acute kidney injury diagnosis defined by KDIGO criteria (Stage 1, 2, 3) during seven days after surgery

SECONDARY OUTCOMES:
Acute kidney injury as defined by AKIN (acute kidney injury network) criteria | within 48 hours after surgery
  Acute kidney injury as defined by AKIN (acute kidney injury network) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea